CLINICAL TRIAL: NCT01030913
Title: B-CLL Subgroups: Maturation Stage and Gene Expression
Brief Title: B-type Chronic Lymphocytic Leukemia (B-CLL) Subgroups: Maturation Stage and Gene Expression
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 04-057
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Cells, Bone Marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia: Chronic Lymphocytic Leukemia

SUMMARY:
B type chronic lymphocytic leukemia (B-CLL) is the most prevalent leukemia in the western world. It is a disease that occurs primarily in aging individuals and occurs more frequently in males than females. Although B-CLL was considered a homogeneous condition, recent studies by our laboratory and others suggest that B-CLL cases can be divided into two subgroups.

These sub-groups can be identified by either the presence or the absence of mutations in antibody genes and/or by the percentage of B-CLL cells expressing a particular protein called CD38. These two sub-groups (unmutated antibody genes high percent CD38 and mutated antibody genes low percentage CD38) follow strikingly clinically different courses. For example, the unmutated/CD38+ group experiences a much more aggressive disease and these patients almost invariably die much sooner than the cases in the other group. In addition, the patients in the mutated CD38+ group require much more chemotherapy than mutatedlCD38-. Finally, surprisingly there is a much higher representation of males in the poor outcome unmutated CD38 group than in the better outcome group. The reasons for these differences in clinical outcome and gender bias are unknown.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,
* Patients must be able to contribute the required amount of blood without compromising their well being,
* Participants must be willing to be contacted again in the future for additional blood drawing.

Exclusion Criteria:

* Patients who are known to be anemic, with a hemoglobin < 8,
* Patients who are known to be infected with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Lymphocytic Leukemia Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 1999-12; Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
differentiating B-CLL cells by the presence or absence of mutations in antibody genes and/or by the percentage of cells expressing CD38 and the difference in clinical disease course and outcome for each group | follow through the clinical disease course for each group

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Chiorazzi, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute for Medical research, Manhasset, New York, United States